CLINICAL TRIAL: NCT05429086
Title: Explore the Advantages of Remimazolam Used on Gastroscopy : A Large Sample, Multicenter, Randomized, Double-blind, Parallel-controlled Clinical Study
Brief Title: Explore the Advantages of Remimazolam Used on Gastroscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Mengchang Yang, Director, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HR7056-IIT
Record Dates: First submitted 2022-06-04; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Induction of Anesthesia
Keywords: remimazolam; propofol
MeSH Terms: interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group remimazolam (Active Comparator): The initial dose of remimazolam was 0.2mg/kg, and the intravenous infusion time was 30s. Within 1 minute (inclusive) of the end of the initial dose: if the subject has achieved sufficient sedation (MOAA/S score ≤3), the gastroscopy will begin; If MOAA/S score > 3 point, additional administration of remimazoalm will be allowed 1 minute after the end of the initial dose. If the MOAA/S score was >3 after 3 consecutive times of addition, sedation failure was determined, and the study was recorded and quit. The drug was given according to clinical needs and the examination was completed. Maintenance of sedation after gastroscopy: In order to maintain a certain degree of sedation after gastroscopy , the evaluator decides when to administer additional drugs.
  remimazolam supplemental administration: the supplemental dose was 2.5 mg , bolus
  Interventions: Drug: Remimazolam
- group propofol (Active Comparator): The initial dose of propofol was 2mg/kg, and the intravenous infusion time was 30s. Within 1 minute (inclusive) of the end of the initial dose: if the subject has achieved sufficient sedation (MOAA/S score ≤3), the gastroscopy will commence. If subjects' MOAA/S score > 3 point, additional administration of propofol will be allowed 1 minute after the end of the initial dose. If the MOAA/S score was >3 after 3 consecutive times of addition, sedation failure was determined, and the study was recorded and quit. The drug was given according to clinical needs and the examination was completed. Maintenance of sedation after gastroscopy: In order to maintain a certain degree of sedation after gastroscopy , the evaluator decides when to administer additional drugs.
  Propofol supplemental administration: the supplemental dose was 0.5mg/kg, bolus.
  Interventions: Drug: Propofol
- group remimazolam combined propofol (Experimental): The initial dose of remimazolam was 0.1 mg/kg, combined propofol 0.5mg/kg, and the infusion time was 30s. Within 1 minute (inclusive) of the end of the initial dose: if the subject has achieved sufficient sedation (MOAA/S score ≤3), the gastroscopy will begin. If subjects' MOAA/S score > 3, additional administration of propofol will be allowed. If the MOAA/S score was >3 after 3 consecutive times of addition, sedation was failure, and the study was recorded and quit. Maintenance of sedation after gastroscopy: In order to maintain a certain degree of sedation after gastroscopy, the evaluator decides when to administer additional drugs.
  supplemental administration: the supplemental dose was remimazolam 2.5 mg,single dose, bolus. There is no permission to use propofol , unless the MOAA/S score still > 3 after five consecutive dosing supplement
  Interventions: Drug: Remimazolam combined propofol

INTERVENTIONS:
Drug: Remimazolam combined propofol — Remimazolam combined propofol
  Arms: group remimazolam combined propofol
Drug: Remimazolam — remimazolam only
  Arms: group remimazolam
Drug: Propofol — propofol only
  Arms: group propofol

SUMMARY:
There are many different types of intravenous anesthetics used in gastroscopy, but each type of drug has its advantages and disadvantages,remimazolam is a novel ultra-short-acting benzodiazepine with rapid onset and recovery, low circulatory depression, and rapid reversal of sedation by flumazenil,remimazolam may be another relatively ideal sedative-hypnotic option for anesthesiologists and gastrointestinal endoscopists. The purpose of this study was to explore whether remimazolam combined with propofol is safer and more effective than remimazolam alone or propofol alone in gastrointestinal endoscopy.

DETAILED DESCRIPTION:
Sedation for gastroscopy is still a topic of debate in the global anesthesia and gastroenterology communities, and the sedation protocols of anesthesiologists and endoscopists vary widely. There are many different types of intravenous anesthetic drugs used in gastroscopy, but each type of drug has its advantages and disadvantages, and the most common protocol in anesthesia practice is an opioid (e.g., fentanyl) combined with a sedative-hypnotic drug (e.g., propofol and midazolam). But these protocols usually have limitations with propofol mainly focusing on respiratory depression and circulatory depression, in which perioperative hypotension should be considered a serious public health problem and should be taken seriously by clinicians, while midazolam has a long onset of action and a long recovery time. Therefore, there is an urgent clinical need for a fast-onset, fast-recovery drug with a high safety profile to solve this current dilemma.

As a new ultra-short-acting benzodiazepine with rapid onset and recovery, low circulatory depression, and rapid reversal of sedation by flumazenil, remimazolam may be another relatively ideal sedative-hypnotic option for anesthesiologists and gastrointestinal endoscopists. The drug was approved for procedural sedation in 2020, and there are many studies on the use of remimazolam versus propofol in gastrointestinal endoscopy sedation. A non-inferiority clinical study of remimazolam tosilate in the upper gastrointestinal tract showed that remimazolam had a sedation success rate no lower than that of propofol, a longer onset of sedation than propofol, but a shorter time to full consciousness than propofol, and a significantly lower incidence of adverse events than propofol. These findings suggest that remimazolam is indeed safer than propofol, but its depth of sedation may be inferior to that of propofol. For clinical workers, it is also essential to have good depth of sedation while ensuring safety. Therefore, considering the above, we hypothesized that the use of remimazolam in combination with propofol in gastrointestinal endoscopy could meet clinical sedation needs and also reduce the incidence of respiratory depression and circulatory depression, which have not been reported. The purpose of this study was to determine whether remimazolam combined with propofol is safer and more effective than remimazolam alone or propofol alone in gastrointestinal endoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are to undergo painless gastroscopy
2. Patients aged 18 - 80 years, regardless of gender
3. 18 < BMI < 30 kg/m2.
4. American Society of Anesthesiologists (ASA) classification of I-III.

Exclusion Criteria:

1. Preoperative hypertensive patients >180/110 mm Hg or hypotensive patients <80/50 mm Hg.
2. Heart rate <50 beats/min.
3. A history of acute inflammation of the respiratory tract that has not been cured within 2 weeks; severe metabolic diseases of the heart, brain, lungs, liver, kidneys and diabetes mellitus; previous heart attack, severe myocardial, ischemia, severe atrioventricular block
4. Those who may have or have had a difficult airway or a history of recovery from abnormal surgical anesthesia
5. Patients with significant electrolyte disturbances such as hyperkalemia
6. Patients with a history of long-term use of immunosuppressive agents such as hormones or adrenal cortical suppression
7. Patients with known allergy to emulsions and opioids
8. Those with combined use of other sedative and analgesic drugs within the preoperative period (including injections, oral and use of related proprietary Chinese medicines)
9. Those suspected of abusing narcotic analgesics or sedatives
10. Those who have neuromuscular system diseases, mental diseases, etc. who do not cooperate and cannot communicate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypotension | Day 1
  20% lower blood pressure than before the drug was administered

SECONDARY OUTCOMES:
Sedation success time | Day 1
  MOAA/S score ≤ 3
Injection pain | Day 1
  the pain score when give the subjects administration
Orientational force score | Day 1
  ask the participants questions to evaluate
Ataxia Scale | Day 1
  teach the participants some motions , then ask them repeat the motions

REFERENCES:
- [Derived] Wei A, Ma S, Dou Y, Wang X, Wu J, Zhou S, Deng Y, Liu X, Li D, Yang M. The safety and efficacy of remimazolam tosylate combined with propofol in upper gastrointestinal endoscopy: A multicenter, randomized clinical trial. PLoS One. 2023 Aug 3;18(8):e0282930. doi: 10.1371/journal.pone.0282930. eCollection 2023. PMID 37535618